CLINICAL TRIAL: NCT01066663
Title: A Phase I/II Study of Pyrimethamine, a STAT3 Inhibitor, for the Treatment of Relapsed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Pyrimethamine for the Treatment of Relapsed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Lymphoma Research Foundation (Other)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 09-421
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2022-12-01 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
Keywords: CLL; SLL; relapsed; pyrimethamine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DL1: Pyrimethamine 12.5 mg (Experimental): Pyrimethamine single daily oral 12.5 mg dose.
  Interventions: Drug: pyrimethamine
- DL2: Pyrimethamine 25 mg (Experimental): Pyrimethamine single daily oral 25 mg dose.
  Interventions: Drug: pyrimethamine
- DL3: Pyrimethamine 50 mg (Experimental): Pyrimethamine single daily oral 50 mg dose.
  Interventions: Drug: pyrimethamine

INTERVENTIONS:
Drug: pyrimethamine — Taken orally once a day
  Other Names: daraprim

SUMMARY:
In this research study we will start by looking for the highest dose of pyrimethamine that can be given safely to CLL patients without severe or unmanageable side effects. This dose will then be used for a larger Phase II study to assess the efficacy of pyrimethamine for the treatment of CLL/SLL. Pyrimethamine is an antibiotic that is used for the treatment of certain infections. Previous research studies have shown that pyrimethamine may target a protein in tumor cells, called STAT3, which may be important for the growth of chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) cells. Pyrimethamine can kill CLL/SLL cells in the laboratory, and we are therefore undertaking this study to assess whether pyrimethamine will result in clinical benefit or tumor responses in CLL in patients.

DETAILED DESCRIPTION:
* Participants will be required to enroll in DFCI Protocol 99-224, the CLL Research Consortium Tissue Bank, and DFCI Protocol 01-206, Tissue and Data Collection for Research Studies in Patients with Hematologic Malignancies, Bone Marrow Disorders, and Normal Donors, or may have blood banked for future use.
* Each treatment cycle lasts 28 days during which time participants will take pyrimethamine orally once per day. Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects, not everyone who participates will receive the same dose of study drug.
* The following tests and procedures will be performed at specific time points during participation in the study: Physical exam, vital signs, blood tests and bone marrow biopsy. The participant's tumor will be assessed by CT scans of the chest, abdomen and pelvis prior to the start of the study and at the end of the 1st, 3rd and 6th months.
* Participants can continue to receive pyrimethamine as long as they do not have side effects and their disease does not worsen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CLL/SLL based on the standard histologic and immunophenotypic criteria described in the WHO classification of lymphoid malignancies, including immunophenotypic confirmation that the tumor cells co-express B cell antigens CD19/20 and CD5. Mantle cell lymphoma should be excluded based on positive staining of the tumor cells for CD23, or the absence of staining of the tumor cells for cyclin D1 or the absence of t(11;14). This diagnosis should be confirmed at a Dana-Farber/Harvard Cancer Center institution within approximately one month after the subject is registered.
* Measurable disease, defined as lymphocytosis > 5,000/uL, or at least one palpable or CT measurable lesion > approximately 1.5cm, or bone marrow involvement > approximately 30%
* Relapsed after at least one prior purine analogue-containing regimen, or at least two non-purine analogue containing regimens
* 18 years of age or older
* Life expectancy of greater than 3 months
* ECOG performance status of 0, 1 or 2
* Normal organ function as outlined in the protocol
* Require treatment based on IWCLL 2008 criteria
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Chemotherapy or radiotherapy within 3 weeks prior to entering the study or those who have not recovered from clinically significant adverse events due to agents administered more than 3 weeks earlier.
* May not be receiving any other study agents
* Known CNS involvement with CLL
* History of allergic reactions or sensitivity to pyrimethamine
* Patients taking folic acid are eligible if the folic acid is discontinued prior to pyrimethamine administration and not taken for the duration of time enrolled on this study
* Prior allogeneic SCT is an exclusion only if the subject has active graft vs. host disease or requires immunosuppression other than a constant stable dose of glucocorticoids
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding women
* HIV-positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2023-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from May 2010 to April 2012
Period: Overall Study
Arm/Group | DL1: Pyrimethamine 12.5 mg | DL2: Pyrimethamine 25 mg | DL3: Pyrimethamine 50 mg
Started | 3 | 3 | 10
Completed | 3 | 3 | 9
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DL1: Pyrimethamine 12.5 mg | DL2: Pyrimethamine 25 mg | DL3: Pyrimethamine 50 mg | Total
Number analyzed (Participants) | 3 | 3 | 10 | 16
Age, Continuous [Median (Full Range); unit: years] | 53 [47 to 79] | 54 [53 to 57] | 60 [31 to 77] | 56 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 5 | 5
  Male | 3 | 3 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 3 | 9 | 14
  Black or African American | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD)
Description: maximum tolerated dose and recommended Phase 2 dose pyrimethamine
Time Frame: Disease were evaluated weekly in 1st 28 days, and every 2 weeks in 2nd cycle then monthly. Median treatment duration is 1.07 months with range 0.23-9.99 months.
Measure: Number; unit: mg
Groups:
- Pyrimethamine Phase 1 (Dose-escalation): Pyrimethamine single daily oral 12.5 mg. 25 mg, or 50 mg dose for dose escalation to determine the MTD
Arm/Group | Pyrimethamine Phase 1 (Dose-escalation)
Number analyzed (Participants) | 16
mg | NA — too few dose limiting toxicities so it is not statistically detectable

2. Primary Outcome: Phase II: Overall Response Rate (ORR)
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Within 10 days of the completion of the cycle required for response evaluation
Population: The phase 2 study were not done and data not collected
Groups:
- Pyrimethamine Phase 2 Dose: Pyrimethamine single daily dose (never went to Phase 2)
Arm/Group | Pyrimethamine Phase 2 Dose
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Grade 3 or Higher Treatment-Related Toxicity
Description: All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAE as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.
Time Frame: as for outcome 1
Measure: Number; unit: number of new cases per 1000 person year
Arm/Group | DL1: Pyrimethamine 12.5 mg | DL2: Pyrimethamine 25 mg | DL3: Pyrimethamine 50 mg
Number analyzed (Participants) | 3 | 3 | 10
number of new cases per 1000 person year | 1 | 5 | 8

4. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease were evaluated weekly in 1st 28 days, and every 2 weeks in 2nd cycle then monthly, and every 3-6 months during the follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DL1: Pyrimethamine 12.5 mg | DL2: Pyrimethamine 25 mg | DL3: Pyrimethamine 50 mg
Number analyzed (Participants) | 3 | 3 | 10
months | 1.116 [0.46 to NA] — Upper confidence interval not statistically reachable | 3.677 [2.791 to NA] — Upper confidence interval not statistically reachable | 0.969 [0.591 to NA] — Upper confidence interval not statistically reachable

ADVERSE EVENTS:
Time Frame: AE were evaluated weekly in 1st 28 days, and every 2 weeks in 2nd cycle then monthly. Median treatment duration is 1.07 months with range 0.23-9.99 months.
Arm/Group | DL1: Pyrimethamine 12.5 mg | DL2: Pyrimethamine 25 mg | DL3: Pyrimethamine 50 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 6/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DL1: Pyrimethamine 12.5 mg (N=3) | DL2: Pyrimethamine 25 mg (N=3) | DL3: Pyrimethamine 50 mg (N=10)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1 | 0
Blood gonadotrophin abnormal (Investigations) | 0 | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 3
Platelet count decreased (Investigations) | 1 | 1 | 3
White blood cell decreased (Investigations) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | DL1: Pyrimethamine 12.5 mg (N=3) | DL2: Pyrimethamine 25 mg (N=3) | DL3: Pyrimethamine 50 mg (N=10)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0/0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 2 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 2 | 9
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 4
Blood bilirubin increased (Investigations) | 1 | 0 | 2
Blood gonadotrophin abnormal (Investigations) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Creatinine increased (Investigations) | 3 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Edema limbs (General disorders) | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 5
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 2
INR increased (Investigations) | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1
Platelet count decreased (Investigations) | 2 | 3 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT01066663/Prot_SAP_000.pdf